CLINICAL TRIAL: NCT05775952
Title: Comparison of Airway Remodeling Mediators Following Experimental Human Rhinovirus Infection in Subjects With Mild to Moderate Asthma and Healthy, Non-asthmatic Control Subjects
Brief Title: Airway Remodeling and Rhinovirus in Asthmatics
Acronym: ARRA
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: ARRA
Record Dates: First submitted 2022-11-17; First posted 2023-03-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Asthma; Respiratory Disease
Keywords: Human Rhinovirus
MeSH Terms: conditions — Asthma; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma Cohort: Subjects with well-controlled, mild-moderate asthma (≥12% post-bronchodilator reversibility or PC20 methacholine <16mg/mL at screening or within past 5 years).
  Subjects will be inoculated with a total dose of 1000 tissue culture-infective dose 50% (TCID50) of rhinovirus (HRV) 39. The inoculum is diluted as appropriate in lactated Ringer's solution and delivered via a two step procedure: 0.25 ml per nostril is administered by pipette while the subject tilts their head back. It is anticipated that subjects will develop mild to moderate symptoms that are transient (lasting 3-7 days) and typically consist of nasal congestion, throat irritation, malaise and increased mucoid secretions. Subjects will record cold symptoms twice daily, using a diary card listing 8 symptoms, each of which are scored 0 to 3 on a basis of severity.
  Subjects will only be inoculated with HRV-39 once at Visit 5.
  Interventions: Biological: HRV-39
- Healthy, Non-asthmatic Cohort: Healthy non-asthmatic control subjects.
  Subjects will be inoculated with a total dose of 1000 tissue culture-infective dose 50% (TCID50) of rhinovirus (HRV) 39. The inoculum is diluted as appropriate in lactated Ringer's solution and delivered via a two step procedure: 0.25 ml per nostril is administered by pipette while the subject tilts their head back. It is anticipated that subjects will develop mild to moderate symptoms that are transient (lasting 3-7 days) and typically consist of nasal congestion, throat irritation, malaise and increased mucoid secretions. Subjects will record cold symptoms twice daily, using a diary card listing 8 symptoms, each of which are scored 0 to 3 on a basis of severity.
  Subjects will only be inoculated with HRV-39 once at Visit 5.
  Interventions: Biological: HRV-39

INTERVENTIONS:
Biological: HRV-39 — We will use a US Food and Drug Administration (FDA) approved Good Manufacturing Practices (GMP)-grade HRV-39 for our proposed study. Use of this GMP-grade HRV-39 viral stock ensures compliance with recent regulatory agency requirements which, beginning in 2001, have mandated that HRV preparations used for human inoculation be made under Good Manufacturing Practices (GMP). This proposed clinical study will allow us to address fundamental questions regarding the nature, kinetics and potential mechanisms of upper and lower airway inflammatory responses in subjects with well-controlled mild-moderate asthma and in healthy, non-asthmatic control subjects; a better understanding of these mechanisms may lead to new paradigms in the treatment of virally-induced airway remodeling and asthma exacerbations.

SUMMARY:
Human rhinovirus is also called the "common cold virus" because it causes at least half of all of the common colds experienced each year. In patients with asthma, getting a rhinovirus infection can cause worsening of asthma symptoms. Although these symptoms are well known, researchers do not fully understand how the virus worsens these asthma symptoms, nor do they really know whether virus infection causes longer term structural changes (often referred to as airway remodeling) in the airways. This study plans to address and answer these questions. Doing so will provide the researchers with a better understanding of how to treat the worsening of asthma that are caused by human rhinovirus infections.

The epithelial cell is the cell that lines the surface of your airways from your nose down to your lungs, and is also the cell type that gets infected by rhinovirus. At present, it is thought that the virus causes symptoms by changing epithelial cell biology in a way that causes airway inflammation. Some of these inflammatory molecules are also thought to cause scarring (remodeling) of the airways, which over time, may lead to a loss of lung function. In order to examine how the virus causes inflammation, many earlier studies have used experimental infection with the virus and have measured various markers of inflammation.

The purpose of this study is to compare the levels of inflammatory and remodeling products in the airways of study participants with mild to moderate asthma and healthy, non-asthmatic subjects after infection with rhinovirus (the common cold virus).

DETAILED DESCRIPTION:
Airway remodeling is a characteristic feature of asthma, and refers to the structural changes that are present in the airways of asthmatic individuals. These changes are considered to be a major contributor to the pathophysiology of the episodic airway dysfunction, termed airway hyperresponsiveness (AHR) that is a hallmark of asthma. The traditional paradigm has, until recently, held that airway remodeling occurs after many years of chronic inflammation. However, more recently, studies have confirmed that remodeling changes are observed in children, in some instances even before the formal diagnosis of asthma is established. Moreover, there is now robust evidence to indicate that children with recurrent human rhinovirus (HRV)-induced wheezing episodes are at significantly increased risk of developing subsequent asthma. This has led us to hypothesize that HRV infections play a role in the development and subsequent continued progression of airway remodeling. In support of this paradigm-shifting hypothesis, we have published novel data, both in vitro and in vivo, establishing that HRV infections up-regulate airway epithelial cell production of several important mediators involved in airway remodeling remodeling processes.

A potential limitation of the in vivo studies reported by us to date is that these have involved healthy, non-asthmatic research participants studied during naturally-acquired HRV infections. Such studies are subject to seasonal variability and are difficult to perform in well-defined study populations, due to uncertainty regarding the onset of infection and the kinetics of subsequent host inflammatory responses. We therefore plan perform a Phase II clinical trial in which we will perform experimental HRV infections in subjects with mild-moderate asthma and in healthy control subjects. This will allow us to accurately study the kinetics of HRV-induced inflammatory and remodeling responses in a well characterized cohort of asthmatic subjects and compare these outcomes to those in a healthy, non-asthmatic control cohort. The primary study outcome will be to determine if alterations in relevant airway remodeling growth factors differ between healthy controls and asthmatic subjects pre- and post-HRV infection. These growth factors will be assessed in bronchoalveolar lavage fluid (BALF) and endobronchial biopsy tissues and correlated with viral titres in both nasal lavage and BALF.

Airway epithelial cells are the primary site of HRV infection, and are the only cell type in which HRV has been detected thus far during in vivo infections. Moreover, there is unequivocal evidence that, following experimental nasal HRV inoculation, virus spreads to infect lower airway epithelial cells, providing a strong biological rationale for the proposed clinical study. HRV only replicate productively in vivo in humans and higher primates and even though rhinoviruses replicate in higher primates (chimpanzees and gibbons), infected animals do not show symptoms. Although two recent publications have reported induction of airway inflammation following exposure of mice to massive doses of unpurified HRV, these responses were transient with little evidence of sustained viral replication. Consequently, we hold the view that HRV only causes relevant infections in vivo in humans and it is for that reason that we continue to focus exclusively on human model systems for all our experimental work. A better understanding of in vivo HRV-induced airway remodeling mediators, and the mechanisms that regulate them, should extend our understanding of the role of HRV infections in the pathogenesis of airway remodeling in asthma.

Clinical studies involving the experimental infection of volunteers with rhinovirus have been conducted for more than 40 years. Challenge pools of rhinovirus for these experiments have generally been produced and safety tested according to guidelines published in 1964 and updated in 1992. The challenge pools produced under these guidelines appeared to be safe. Multiple studies have been conducted over this 40-year period in several countries. Dr. Proud has over 20 years of experience in conducting experimental HRV infection protocols. In the 40 years of such studies, it is reasonable to estimate that some 10,000 volunteers have been challenged worldwide to date, and no serious complications attributable to the viral infection have been detected. Moreover, nearly a dozen experimental HRV infection studies have been done in subjects with mild-moderate asthma over the past decade without serious complications. While these studies have contributed substantially to our understanding of rhinovirus-induced asthma symptoms, as well as of host inflammatory and antiviral responses, none have yet looked at the effects of experimental HRV infection on indices of airway remodeling.

Therefore, as a natural extension of our current research program and, in keeping with our expertise in HRV-related research, we now plan to perform this experimental rhinovirus infection study. We plan to use a US Food and Drug Administration (FDA) approved Good Manufacturing Practices (GMP)-grade HRV-39 (a gift from Dr. Ronald B. Turner, University of Virginia) for our proposed study. Use of this GMP-grade HRV-39 viral stock ensures compliance with recent regulatory agency requirements which, beginning in 2001, have mandated that HRV preparations used for human inoculation be made under Good Manufacturing Practices (GMP). This proposed clinical study will allow us to address fundamental questions regarding the nature, kinetics and potential mechanisms of upper and lower airway inflammatory responses in subjects with well-controlled mild-moderate asthma and in healthy, non-asthmatic control subjects; a better understanding of these mechanisms may lead to new paradigms in the treatment of virally-induced airway remodeling and asthma exacerbations.

ELIGIBILITY:
Asthma Cohort

Inclusion Criteria:

* Male or female volunteers with intermittent or persistent mild to moderate allergic asthma, as defined by GINA guidelines.
* Between ≥18 and ≤ 65 years of age
* Objective evidence of variable airflow limitation (≥12% and at least 200mL post-bronchodilator reversibility from baseline) and airway hyperresponsiveness (PC20 methacholine <16mg/mL) at screening or within past 5 years
* Spirometry at baseline shows FEV1 ≥ 60% of predicted; FEV1/FVC ≥ 0.40
* Atopic, as evidenced by positive skin prick tests to ≥1 common aero-allergen, where positive is defined by a wheal of ≥2 mm greater than the negative control
* Not be exposed to sensitizing seasonal allergens for at least 4 weeks before visit 2
* Asthma symptoms controlled by either inhaled beta 2-agonists alone, or by low or moderate dose (≤800 μg of budesonide or equivalent per day) inhaled corticosteroid (ICS) administered either as monotherapy or in a fixed-dose combination with a long-acting beta 2-agonist (LABA)
* Be a non-smoker for ≥1 year and have a lifetime ≤ 10 pack-year smoking history of smoking
* In good general health (other than asthma) without clinically significant medical history of other comorbidities, and a BMI of ≤ 35 kg/m2.

Healthy, Non-asthmatic Cohort

Inclusion Criteria:

* Male or female volunteers in good general health, without clinically significant medical history and a BMI of ≤ 35 kg/m2
* Between ≥18 and ≤ 65 years of age
* Non-asthmatic, as defined by history and normal spirometry (FEV1 ≥80% predicted; FEV1/FVC ≥ 0.75)
* Normal airway responsiveness (PC20 methacholine not detected at, or less than, 16 mg/mL)
* Non-atopic, as determined by skin prick tests to common aero-allergens, where a positive test is defined as a wheal of ≥2 mm greater than the negative control.
* Be a non-smoker for ≥1 year and have a lifetime ≤ 10 pack-year smoking history of smoking
* Willing to participate in study and be able to provide written consent prior to starting the study.

Exclusion Criteria (both cohorts):

* Presence of neutralizing antibodies to HRV-39
* Current pregnancy or positive urine pregnancy test at screening
* Use of any of the following medications: antihistamines, leukotriene antagonists, inhaled anticholinergics, non-steroidal anti-inflammatories, antibiotics, and over the counter 'cold' and influenza remedies, in preceding 4 weeks prior to visit 2.
* Current acute or chronic illness (including infection) or recent recovery (within 4 weeks of visit 3) from acute illness which could, in the opinion of the Investigator, alter inflammatory responses (e.g., flu, cold or other respiratory infection, etc.).
* Autoimmune disease or immunodeficiency
* Any other significant concomitant medical issue, or findings on physical examination or medical history that, in the opinion of the study physician, may pose additional risks from participation in the study (including undergoing bronchoscopy), or which may impact the quality or interpretation of the data obtained from the study.
* Inability or unwillingness of a potentially eligible study participant to give written informed consent.
* Unable or unwilling to adhere to protocol-defined study visit schedule and/or other protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All potentially eligible study subjects will be screened for the presence of neutralizing serum antibodies to HRV-39 and only those subjects who are seronegative for HRV-39 will be included in either of the study cohorts:
  1. Twelve non-smoking subjects with mild-moderate atopic asthma, aged 18-65 years, will be asked to volunteer for the study.
  2. Twelve healthy non-smoking, non-allergic, non-asthmatic subjects, aged 18-65 years, will be asked to volunteer for the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2011-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The change between pre- and post-rhinoviral infection. | Baseline (Visit 1) to Week 8 (Visit 11).
  Experimental rhinoviral infection will be confirmed by detection of viral shedding in nasal lavage fluids using conventional viral titre assay using MRC-5 fibroblasts, RT-PCR for HRV 39 viral RNA and standard viral titer assays, and/or by a 4-fold increase in HRV-39 neutralizing serum antibody titre 4 weeks after infection.
Change of protein levels. | Screening (Visit 4; Week 2) to infectious phase (Visit 9; Week 4).
  Immunohistochemistry will be performed on bronchial biopsies to identify the following cells: total leukocytes (CD45+), T-lymphocytes (CD3+), T-lymphocyte subsets (CD4+ and CD8+), B-lymphocytes (CD20+), neutrophils (anti-neutrophil elastase), macrophages (CD68+), mast cells (anti-tryptase, AA1), myofibroblasts (α-smooth muscle actin) and blood vessels (CD34+).
The change in the lower airway secretions and tissues for selected airway remodeling mediators. | Screening (Visit 4; Week 2) to infectious phase (Visit 9; Week 4).
  Airway remodeling mediators including matrix metalloproteinase (MMP)-9, amphiregulin, vascular endothelial growth factor (VEGF) and activin A will be assess from bronchial lavage and biopsy samples.

SECONDARY OUTCOMES:
Quantitative changes | Screening (Visit 4; Week 2) to infectious phase (Visit 9; Week 4).
  Quantitative changes in gene expression, expressed in absolute units (e.g. attograms) between groups in lower airway secretions and tissues, as well as nasal scrapings, for selected airway remodeling mediator genes, including MMP-9, amphiregulin, VEGF and activin A.
  Quantitative changes in gene expression, expressed in absolute units (e.g. attograms) between groups in lower airway secretions and tissues, as well as nasal scrapings, for selected novel airway remodeling mediator genes, identified by us to be unregulated by HRV infection on recent gene array studies
Number of airway myofibroblasts | Screening (Visit 4; Week 2) to infectious phase (Visit 9; Week 4).
  Changes in the number of airway myofibroblasts in bronchial biopsies following HRV-39 infection. We have recently reported a dramatic increase in the numbers of airway myofibroblasts 24 h post allergen challenge, and will now determine if similar changes occur in response to HRV infection.
Changes in symptom scores - asthma control questionnaire (ACQ) | Baseline (Visit 1) to Week 8 (Visit 11).
  Changes in symptom scores (asthma control questionnaire (ACQ), measured on a scale from 1-6
Changes in cold symptom questionnaire | Baseline (Visit 1) to Week 8 (Visit 11).
  cold symptom questionnaire, measured on a scale of 1-6
Changes in viral titres | Baseline (Visit 1) to Week 8 (Visit 11).
  Viral titres (measured with TCDI50)
Changes in spirometry | Baseline (Visit 1) to Week 8 (Visit 11).
  spirometry (measured by FEV1/FVC; Asthma cohort, FEV1 ≥ 60% of predicted; FEV1/FVC ≥ 0.40; Non-asthmatic, FEV1 ≥80% predicted; FEV1/FVC ≥ 0.75)
Changes in airway responsiveness | Baseline (Visit 1) to Week 8 (Visit 11).
  Airway responsiveness (measured by methacholine challenge)
Changes in FeNO levels | Baseline (Visit 1) to Week 8 (Visit 11).
  FeNO levels (measured in ppb)
Gene expression and protein levels | Baseline (Visit 1) to Week 8 (Visit 11).
  The correlation of gene expression and protein levels of selected mediators with viral titer, symptom scores and the numbers of inflammatory cells in the upper and lower airways.
Quantitation of inflammatory cells in the lower airways, assessed in BALF and bronchial biopsies. | Screening (Visit 4; Week 2) to infectious phase (Visit 9; Week 4).
  Quantitation of inflammatory cells in the lower airways, assessed in BALF and bronchial biopsies using FACS, H & E staining to determine the adequacy and general morphology of the sample, Masson's Trichome stain and Picrosirius Red to demonstrate the presence of extracellular-matrix, and periodic acid Schiff (PAS) to demonstrate the presence of mucin within goblet cells.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leigh R, Oyelusi W, Wiehler S, Koetzler R, Zaheer RS, Newton R, Proud D. Human rhinovirus infection enhances airway epithelial cell production of growth factors involved in airway remodeling. J Allergy Clin Immunol. 2008 May;121(5):1238-1245.e4. doi: 10.1016/j.jaci.2008.01.067. Epub 2008 Mar 19. PMID 18355907
- [Background] Tacon CE, Wiehler S, Holden NS, Newton R, Proud D, Leigh R. Human rhinovirus infection up-regulates MMP-9 production in airway epithelial cells via NF-kappaB. Am J Respir Cell Mol Biol. 2010 Aug;43(2):201-9. doi: 10.1165/rcmb.2009-0216OC. Epub 2009 Sep 25. PMID 19783786
- [Background] Turner RB, Hendley JO, Gwaltney JM Jr. Shedding of infected ciliated epithelial cells in rhinovirus colds. J Infect Dis. 1982 Jun;145(6):849-53. doi: 10.1093/infdis/145.6.849. PMID 6282984
- [Background] Bardin PG, Johnston SL, Sanderson G, Robinson BS, Pickett MA, Fraenkel DJ, Holgate ST. Detection of rhinovirus infection of the nasal mucosa by oligonucleotide in situ hybridization. Am J Respir Cell Mol Biol. 1994 Feb;10(2):207-13. doi: 10.1165/ajrcmb.10.2.8110476.
- [Background] Arruda E, Boyle TR, Winther B, Pevear DC, Gwaltney JM Jr, Hayden FG. Localization of human rhinovirus replication in the upper respiratory tract by in situ hybridization. J Infect Dis. 1995 May;171(5):1329-33. doi: 10.1093/infdis/171.5.1329. PMID 7751712
- [Background] Papadopoulos NG, Bates PJ, Bardin PG, Papi A, Leir SH, Fraenkel DJ, Meyer J, Lackie PM, Sanderson G, Holgate ST, Johnston SL. Rhinoviruses infect the lower airways. J Infect Dis. 2000 Jun;181(6):1875-84. doi: 10.1086/315513. Epub 2000 Jun 5. PMID 10837165
- [Background] Mosser AG, Vrtis R, Burchell L, Lee WM, Dick CR, Weisshaar E, Bock D, Swenson CA, Cornwell RD, Meyer KC, Jarjour NN, Busse WW, Gern JE. Quantitative and qualitative analysis of rhinovirus infection in bronchial tissues. Am J Respir Crit Care Med. 2005 Mar 15;171(6):645-51. doi: 10.1164/rccm.200407-970OC. Epub 2004 Dec 10. PMID 15591468
- [Background] Dick EC. Experimental infections of chimpanzees with human rhinovirus types 14 and 43. Proc Soc Exp Biol Med. 1968 Apr;127(4):1079-81. doi: 10.3181/00379727-127-32875. No abstract available. PMID 4297694
- [Background] Pinto CA, Haff RF. Experimental infection of gibbons with rhinovirus. Nature. 1969 Dec 27;224(5226):1310-1. doi: 10.1038/2241310a0. No abstract available. PMID 4311662
- [Background] Bartlett NW, Walton RP, Edwards MR, Aniscenko J, Caramori G, Zhu J, Glanville N, Choy KJ, Jourdan P, Burnet J, Tuthill TJ, Pedrick MS, Hurle MJ, Plumpton C, Sharp NA, Bussell JN, Swallow DM, Schwarze J, Guy B, Almond JW, Jeffery PK, Lloyd CM, Papi A, Killington RA, Rowlands DJ, Blair ED, Clarke NJ, Johnston SL. Mouse models of rhinovirus-induced disease and exacerbation of allergic airway inflammation. Nat Med. 2008 Feb;14(2):199-204. doi: 10.1038/nm1713. Epub 2008 Feb 3. PMID 18246079
- [Background] Newcomb DC, Sajjan US, Nagarkar DR, Wang Q, Nanua S, Zhou Y, McHenry CL, Hennrick KT, Tsai WC, Bentley JK, Lukacs NW, Johnston SL, Hershenson MB. Human rhinovirus 1B exposure induces phosphatidylinositol 3-kinase-dependent airway inflammation in mice. Am J Respir Crit Care Med. 2008 May 15;177(10):1111-21. doi: 10.1164/rccm.200708-1243OC. Epub 2008 Feb 14. PMID 18276942
- [Background] KNIGHT V. THE USE OF VOLUNTEERS IN MEDICAL VIROLOGY. Prog Med Virol. 1964;6:1-26. No abstract available. PMID 14310573
- [Background] Gwaltney JM Jr, Hendley O, Hayden FG, McIntosh K, Hollinger FB, Melnick JL, Turner RB. Updated recommendations for safety-testing of viral inocula used in volunteer experiments on rhinovirus colds. Prog Med Virol. 1992;39:256-63. No abstract available. PMID 1317600
- [Background] Naclerio RM, Proud D, Lichtenstein LM, Kagey-Sobotka A, Hendley JO, Sorrentino J, Gwaltney JM. Kinins are generated during experimental rhinovirus colds. J Infect Dis. 1988 Jan;157(1):133-42. doi: 10.1093/infdis/157.1.133. PMID 2447198
- [Background] Proud D, Gwaltney JM Jr, Hendley JO, Dinarello CA, Gillis S, Schleimer RP. Increased levels of interleukin-1 are detected in nasal secretions of volunteers during experimental rhinovirus colds. J Infect Dis. 1994 May;169(5):1007-13. doi: 10.1093/infdis/169.5.1007. PMID 8169385
- [Background] Spurrell JC, Wiehler S, Zaheer RS, Sanders SP, Proud D. Human airway epithelial cells produce IP-10 (CXCL10) in vitro and in vivo upon rhinovirus infection. Am J Physiol Lung Cell Mol Physiol. 2005 Jul;289(1):L85-95. doi: 10.1152/ajplung.00397.2004. Epub 2005 Mar 11. PMID 15764644
- [Background] Proud D, Turner RB, Winther B, Wiehler S, Tiesman JP, Reichling TD, Juhlin KD, Fulmer AW, Ho BY, Walanski AA, Poore CL, Mizoguchi H, Jump L, Moore ML, Zukowski CK, Clymer JW. Gene expression profiles during in vivo human rhinovirus infection: insights into the host response. Am J Respir Crit Care Med. 2008 Nov 1;178(9):962-8. doi: 10.1164/rccm.200805-670OC. Epub 2008 Jul 24. PMID 18658112
- [Background] Grunberg K, Kuijpers EA, de Klerk EP, de Gouw HW, Kroes AC, Dick EC, Sterk PJ. Effects of experimental rhinovirus 16 infection on airway hyperresponsiveness to bradykinin in asthmatic subjects in vivo. Am J Respir Crit Care Med. 1997 Mar;155(3):833-8. doi: 10.1164/ajrccm.155.3.9117013.
- [Background] Grunberg K, Timmers MC, Smits HH, de Klerk EP, Dick EC, Spaan WJ, Hiemstra PS, Sterk PJ. Effect of experimental rhinovirus 16 colds on airway hyperresponsiveness to histamine and interleukin-8 in nasal lavage in asthmatic subjects in vivo. Clin Exp Allergy. 1997 Jan;27(1):36-45. doi: 10.1111/j.1365-2222.1997.tb00670.x. PMID 9117878
- [Background] Grunberg K, Smits HH, Timmers MC, de Klerk EP, Dolhain RJ, Dick EC, Hiemstra PS, Sterk PJ. Experimental rhinovirus 16 infection. Effects on cell differentials and soluble markers in sputum in asthmatic subjects. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):609-16. doi: 10.1164/ajrccm.156.2.9610079. PMID 9279247
- [Background] Grunberg K, Timmers MC, de Klerk EP, Dick EC, Sterk PJ. Experimental rhinovirus 16 infection causes variable airway obstruction in subjects with atopic asthma. Am J Respir Crit Care Med. 1999 Oct;160(4):1375-80. doi: 10.1164/ajrccm.160.4.9810083. PMID 10508832
- [Background] Gern JE, Vrtis R, Grindle KA, Swenson C, Busse WW. Relationship of upper and lower airway cytokines to outcome of experimental rhinovirus infection. Am J Respir Crit Care Med. 2000 Dec;162(6):2226-31. doi: 10.1164/ajrccm.162.6.2003019. PMID 11112143
- [Background] Grunberg K, Sharon RF, Hiltermann TJ, Brahim JJ, Dick EC, Sterk PJ, Van Krieken JH. Experimental rhinovirus 16 infection increases intercellular adhesion molecule-1 expression in bronchial epithelium of asthmatics regardless of inhaled steroid treatment. Clin Exp Allergy. 2000 Jul;30(7):1015-23. doi: 10.1046/j.1365-2222.2000.00854.x. PMID 10848925
- [Background] Grunberg K, Sharon RF, Sont JK, In 't Veen JC, Van Schadewijk WA, De Klerk EP, Dick CR, Van Krieken JH, Sterk PJ. Rhinovirus-induced airway inflammation in asthma: effect of treatment with inhaled corticosteroids before and during experimental infection. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 1):1816-22. doi: 10.1164/ajrccm.164.10.2102118. PMID 11734429
- [Background] de Kluijver J, Evertse CE, Sont JK, Schrumpf JA, van Zeijl-van der Ham CJ, Dick CR, Rabe KF, Hiemstra PS, Sterk PJ. Are rhinovirus-induced airway responses in asthma aggravated by chronic allergen exposure? Am J Respir Crit Care Med. 2003 Nov 15;168(10):1174-80. doi: 10.1164/rccm.200212-1520OC. Epub 2003 Jul 31. PMID 12893645
- [Background] Message SD, Laza-Stanca V, Mallia P, Parker HL, Zhu J, Kebadze T, Contoli M, Sanderson G, Kon OM, Papi A, Jeffery PK, Stanciu LA, Johnston SL. Rhinovirus-induced lower respiratory illness is increased in asthma and related to virus load and Th1/2 cytokine and IL-10 production. Proc Natl Acad Sci U S A. 2008 Sep 9;105(36):13562-7. doi: 10.1073/pnas.0804181105. Epub 2008 Sep 3. PMID 18768794
- [Background] DeMore JP, Weisshaar EH, Vrtis RF, Swenson CA, Evans MD, Morin A, Hazel E, Bork JA, Kakumanu S, Sorkness R, Busse WW, Gern JE. Similar colds in subjects with allergic asthma and nonatopic subjects after inoculation with rhinovirus-16. J Allergy Clin Immunol. 2009 Aug;124(2):245-52, 252.e1-3. doi: 10.1016/j.jaci.2009.05.030. Epub 2009 Jul 12. PMID 19596142
- [Background] Bateman ED, Hurd SS, Barnes PJ, Bousquet J, Drazen JM, FitzGerald JM, Gibson P, Ohta K, O'Byrne P, Pedersen SE, Pizzichini E, Sullivan SD, Wenzel SE, Zar HJ. Global strategy for asthma management and prevention: GINA executive summary. Eur Respir J. 2008 Jan;31(1):143-78. doi: 10.1183/09031936.00138707. PMID 18166595
- [Background] Kelly MM, O'Connor TM, Leigh R, Otis J, Gwozd C, Gauvreau GM, Gauldie J, O'Byrne PM. Effects of budesonide and formoterol on allergen-induced airway responses, inflammation, and airway remodeling in asthma. J Allergy Clin Immunol. 2010 Feb;125(2):349-356.e13. doi: 10.1016/j.jaci.2009.09.011. Epub 2009 Dec 6. PMID 19969339
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Recommendations for standardized procedures for the on-line and off-line measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide in adults and children-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 1999 Dec;160(6):2104-17. doi: 10.1164/ajrccm.160.6.ats8-99. No abstract available. PMID 10588636
- [Background] Workshop summary and guidelines: investigative use of bronchoscopy, lavage, and bronchial biopsies in asthma and other airway diseases. J Allergy Clin Immunol. 1991 Nov;88(5):808-14. doi: 10.1016/0091-6749(91)90189-u. No abstract available. PMID 1955640
- [Background] Jeffery P, Holgate S, Wenzel S; Endobronchial Biopsy Workshop. Methods for the assessment of endobronchial biopsies in clinical research: application to studies of pathogenesis and the effects of treatment. Am J Respir Crit Care Med. 2003 Sep 15;168(6 Pt 2):S1-17. doi: 10.1164/rccm.200202-150WS. No abstract available. PMID 14555461
- [Background] Busse WW, Wanner A, Adams K, Reynolds HY, Castro M, Chowdhury B, Kraft M, Levine RJ, Peters SP, Sullivan EJ. Investigative bronchoprovocation and bronchoscopy in airway diseases. Am J Respir Crit Care Med. 2005 Oct 1;172(7):807-16. doi: 10.1164/rccm.200407-966WS. Epub 2005 Jul 14. PMID 16020805